CLINICAL TRIAL: NCT02776332
Title: A Randomized Controlled Trial Comparing The Effect Of Duration Of Manual Expression And Breastfeeding Self-efficacy On Milk Volumes In Mothers Of Premature Infants
Brief Title: The Merit Study (Manual Expression pRemature InfanTs)
Acronym: MERIT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: St. Louis Children's Hospital (Other)
Responsible Party: Principal Investigator, Lisa Steurer PhD (c), RN, CPNP-PC, CLC, APN Professional Practice & Systems, St. Louis Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16-052
Record Dates: First submitted 2016-05-12; First posted 2016-05-18 (Estimated); Last update posted 2018-09-06 (Actual); Status verified 2018-09

CONDITIONS: Breast Milk Expression
Keywords: breastfeeding; premature infants; manual expression
MeSH Terms: conditions — Breast Milk Expression; Breast Feeding; Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 3 day group (Active Comparator): Manual expression for 3 days after delivery Breastfeeding log for 14 days after delivery Video of manual expression for teaching and reinforcement Complete breastfeeding self-efficacy scale at 1 day and 14 days after delivery
  Interventions: Procedure: Manual Expression of Breastmilk
- 7 day group (Active Comparator): The 7 day group will manually express for 7 days after delivery. Breastfeeding log for 14 days after delivery Video of manual expression for teaching and reinforcement Complete breastfeeding self-efficacy scale at 1 day and 14 days after delivery follow up phone call at 5 days to encourage continued manual expression
  Interventions: Procedure: Manual Expression of Breastmilk

INTERVENTIONS:
Procedure: Manual Expression of Breastmilk — Breastfeeding log for 14 days after delivery Video of manual expression for teaching and reinforcement Complete breastfeeding self-efficacy scale at 1 day and 14 days after delivery

SUMMARY:
The purpose of this study is to determine how the duration of manual expression affects milk volumes and levels of breastfeeding self-efficacy in mothers of premature infants.

The specific aims of this study are to determine if the duration of manual expression in mothers of premature infants will result in: (a) an increase in breastfeeding self-efficacy (b) a difference in milk volume and (c) a correlation between breastfeeding self-efficacy and milk volume.

DETAILED DESCRIPTION:
Manual Expression of Breast Milk One of the major contributing factors for the cessation of breast feeding in the premature population of infants is decreased milk production. Because most premature infants are unable to initially feed at the breast, artificial methods to maintain milk supply such as manual and electric pump expression have been explored.

Studies by Flaherman et al. and Slusher et al. both used a randomized design to address manual versus pump expression and its effect on milk volume. Flaherman et al. studied a population of 68 full-term infants feeding poorly at the breast for two months after delivery in a United States academic medical center and randomized the mother to either manual expression or electric pump expression. Slusher et al. allocated mothers of 65 premature infants admitted to an African special care nursery to manual expression, manual powered pedal pump or an electric pump for six-ten days after delivery. Both studies found the electric pump to yield higher volumes of milk than manual expression. Slusher et al. found a statistically significant increase in milk volume with the electric pump when compared to manual expression (p<0.01). No mean differences in demographics between the three groups were found. Flaherman et al. also reported higher milk volumes with the electric pump but the comparison failed to reach statistical significance (p=0.07). Although failing to reach statistical significance on milk volume, Flaherman, followed participants for two months and reported higher rates of continued breastfeeding among the mothers who had initially used hand expression (p=0.02). In addition, Flaherman measured self -efficacy using the Breastfeeding Self-Efficacy Scale-Short Form (BSES-SF) at baseline, one week, one moth and two months after delivery. However, there were no significant differences between the groups for breastfeeding self-efficacy.

Two studies investigated a combination of manual and electric pump expression. Morton combined hand expression and electric pumping whereas Ohyama used manual expression or electric pump expression. In the study by Morton) a prospective observational design was used to examine milk production for eight weeks after delivery for mothers who were instructed to use an electric pump and manually express as much as possible in the first three days post-partum with no particular sequencing. In this sample of 67 mothers of premature infants, Morton was able to find an increased milk production at two weeks for those mothers that hand expressed greater than five times a day (p<0.05). Ohyama also studied mothers of premature infants in a Japanese neonatal intensive care unit using a crossover design that studied a combination of manual and electric pump expression techniques. The mothers were sequentially allocated to either manual or electric pump expression and then alternated the method until seven sessions had been completed for each method. Net milk yield was significantly higher with manual expression (p<0.05) as compared to pump expression in the first 48 hours after delivery. Both of these studies support the potential benefit of manual expression for early removal of colostrum prior to the onset of mature milk.

A pilot feasibility study using a combined sequence of manual and pump expression intervention for the first three days after delivery was conducted on the mothers of premature infants whose infants were hospitalized in a NICU in the proposed study population and setting. Mothers of premature infants (n=6) were asked by staff nurses in the intra-partum and post-partum units to perform manual expression prior to electric pump expression for the first three days after delivery and record milk volumes on a breastfeeding log for three weeks after delivery. Women who had not begun an initial expression within six hours after delivery were initially excluded, based on previous literature that states the longer the delay in time from delivery to expression can serve as an important variable in overall milk production. Due to the infeasibility of the women being able to begin their first pumping session within six hours of delivery due to complications of delivery or other logistical issues within the healthcare setting, the inclusion criteria for recruitment was extended from six hours to 24 hours after delivery. The intervention of manual expression was able to be delivered on all of the mothers in the study thus providing important information on the feasibility of teaching this intervention in this population of mothers. However, because only half of the mothers in the study were able to complete the log, revisions in the amount and duration of study variables for the larger study have been considered.

Limitations of Previous Studies on Manual Expression Of the studies reviewed, only three addressed premature infants and only two were randomized trials thus causation is difficult to establish. There was conflicting evidence whether electric pump expression or manual expression yielded higher milk volumes and a standard sequencing method was not always employed in the research design. All of the studies reported relatively low sample sizes and failed to mention the use of a power analysis which can lead to a Type I error. Most of the studies were focused on physiological outcomes as the primary measure and did not incorporate a theoretical framework. The studies were based on the physiological theory that early and frequent pump expression after delivery is essential to maintain milk supply in mothers who may be separated from their infants or when infants are feeding poorly.

Despite the mixed results of previous studies it is becoming standard practice for many hospitals to instruct all mothers on manual expression as a result of the recommendation of the Baby-Friendly Hospital Initiative (BFHI). The BFHI is a global initiative endorsed by WHO and the United Nations Children's Fund (UNICEF) whose primary goal is to assist all mothers in being able to successfully initiate and sustain breastfeeding. The BFHI recognizes hospitals that are successful in meeting their guidelines for breastfeeding quality and outcomes. The number of U.S. hospitals applying for the BFHI certification has increased since 2010 when the U.S. Department of Health and Human Services incorporated the practices promoted into federal goals. As part of the BFHI global criteria, 80% of mothers need to report that they have been taught how to hand express their milk for both mothers feeding at the breast and for those mothers who are separated from their babies. The duration of manual expression was not defined by the BFHI and previous studies incorporating manual expression have not measured how many days of manual expression may be optimal. Of the studies reviewed that incorporated manual expression as an independent variable, most were not in combination with electric pump expression. The duration of manual expression varied across all studies; anywhere from three to eight days after delivery.

As previously discussed, lactogenesis II is marked by the onset of copious milk secretion after birth and the delivery of the placenta and occurs anywhere from two to eight days postpartum. Due to the variability of when mature milk is created, the timing of the colostrum period may vary per individual. Comparing the duration of manual expression may reveal insights into the optimal timing of this expression technique for mothers of premature infants. No studies reviewed focused on the duration of manual expression as an independent variable. This study will be the first to focus on the duration of manual expression as the primary variable of interest.

ELIGIBILITY:
Inclusion Criteria:

* Participant delivered premature infant (23-34 weeks gestation)
* Intention to breastfeed
* Infant admitted to NICU

Exclusion Criteria:

* Premature infant <23 or > 34 weeks gestation
* Non-English speaking
* Mother critically ill
* History of breast augmentation surgery
* Time lapse of > 24 hours since delivery to first expression of breast milk

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Estimated)
Dates: Start 2016-05-26 (Actual); Primary Completion 2018-12-31 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
Milk Volume | up to 14 days
  Milk volume at each pumping session from day 1-day 14 after delivery

SECONDARY OUTCOMES:
Level of breastfeeding self-efficacy | Day 1 and Day 14
  Baseline and repeated breastfeeding self-efficacy scale (BSES-SF)

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia Russell, PhD, Study Chair — Univeristy of Missouri Kansas City
Locations (1):
- Barnes Jewish Hospital, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dennis CL. The breastfeeding self-efficacy scale: psychometric assessment of the short form. J Obstet Gynecol Neonatal Nurs. 2003 Nov-Dec;32(6):734-44. doi: 10.1177/0884217503258459. PMID 14649593
- [Background] Flaherman VJ, Gay B, Scott C, Avins A, Lee KA, Newman TB. Randomised trial comparing hand expression with breast pumping for mothers of term newborns feeding poorly. Arch Dis Child Fetal Neonatal Ed. 2012 Jan;97(1):F18-23. doi: 10.1136/adc.2010.209213. Epub 2011 Jul 11. PMID 21747129
- [Background] Hill PD, Aldag JC, Zinaman M, Chatterton RT. Predictors of preterm infant feeding methods and perceived insufficient milk supply at week 12 postpartum. J Hum Lact. 2007 Feb;23(1):32-8; quiz 39-43. doi: 10.1177/0890334406297277. PMID 17293549
- [Background] Hill PD, Aldag JC, Chatterton RT, Zinaman M. Primary and secondary mediators' influence on milk output in lactating mothers of preterm and term infants. J Hum Lact. 2005 May;21(2):138-50. doi: 10.1177/0890334405275403. PMID 15886340
- [Background] Morton J, Hall JY, Wong RJ, Thairu L, Benitz WE, Rhine WD. Combining hand techniques with electric pumping increases milk production in mothers of preterm infants. J Perinatol. 2009 Nov;29(11):757-64. doi: 10.1038/jp.2009.87. Epub 2009 Jul 2. PMID 19571815
- [Background] Murase M, Nommsen-Rivers L, Morrow AL, Hatsuno M, Mizuno K, Taki M, Miyazawa T, Nakano Y, Aizawa M, Itabashi K. Predictors of low milk volume among mothers who delivered preterm. J Hum Lact. 2014 Nov;30(4):425-35. doi: 10.1177/0890334414543951. Epub 2014 Jul 25. PMID 25063573
- [Background] Ohyama M, Watabe H, Hayasaka Y. Manual expression and electric breast pumping in the first 48 h after delivery. Pediatr Int. 2010 Feb;52(1):39-43. doi: 10.1111/j.1442-200X.2009.02910.x. Epub 2009 Jun 11. PMID 19519669
- [Background] Slusher T, Slusher IL, Biomdo M, Bode-Thomas F, Curtis BA, Meier P. Electric breast pump use increases maternal milk volume in African nurseries. J Trop Pediatr. 2007 Apr;53(2):125-30. doi: 10.1093/tropej/fml066. PMID 17409102
- [Background] Sisk P, Quandt S, Parson N, Tucker J. Breast milk expression and maintenance in mothers of very low birth weight infants: supports and barriers. J Hum Lact. 2010 Nov;26(4):368-75. doi: 10.1177/0890334410371211. Epub 2010 Oct 7. PMID 20930219